CLINICAL TRIAL: NCT02872103
Title: A Phase III, Randomized, Multi-Centre, Double-Blind, Placebo Controlled Clinical Trial of F-627 in Women With Breast Cancer Receiving Myelotoxic Chemotherapy
Brief Title: Placebo-controlled Trial of F-627 in Women With Breast Cancer Receiving Myelotoxic Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EVIVE Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GC-627-04
Record Dates: First submitted 2016-08-08; First posted 2016-08-19 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Neutropenia
MeSH Terms: conditions — Breast Neoplasms; Neutropenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- F-627 (Experimental): F-627, 20 mg fixed dose pre-filled syringe, dosed Day 2 of each of 4 chemotherapy cycles.
  Interventions: Drug: F-627
- Placebo (Placebo Comparator): Placebo, pre-filled syringe administered Day 2 of the first chemotherapy cycle; and F-627, 20 mg fixed dose pre-filled syringe administered Day 2 of each of the following 3 chemotherapy cycles.
  Interventions: Drug: F-627; Drug: Placebo

INTERVENTIONS:
Drug: F-627 — F-627 subcutaneous injection on Day 2 of TA chemotherapy cycles. TA chemotherapy treatments are part of standard-of-care and not the study
Drug: Placebo — Placebo subcutaneous injection on Day 2 of the first TA chemotherapy cycle. TA chemotherapy treatments are part of standard-of-care and not the study.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind and placebo controlled phase 3 study to evaluate the efficacy and safety of F-627 in women with stage II-IV breast cancer receiving chemotherapy treatment.

DETAILED DESCRIPTION:
This is a randomized, multi-center, single dose, double-blind, placebo controlled phase III study of the efficacy and safety of once-per-cycle of F-627 in women with stage II-IV breast cancer who are receiving myelotoxic TA chemotherapy treatment (Taxotere (docetaxel) + Adriamycin(doxorubicin)). F-627 is designed to treat neutropenia, an abnormally low number of neutrophils (a type of white blood cell) in the blood. Neutropenia is often seen in cancer patients receiving myelotoxic chemotherapy.

The primary objective of this study is to evaluate the efficacy and safety of single fixed dose of F-627 in breast cancer patients experiencing myelotoxic chemotherapy in comparison to placebo. F-627 or placebo is to be administered subcutaneously 24 hours after chemotherapy in each 21-day cycle of chemotherapy treatment (up to 4 cycles). Patients randomized to placebo arm will receive F-627 except in cycle 1. The primary endpoint will be the duration of grade 4 (severe) neutropenia - the number of days in which the patient has had an absolute neutrophil count (ANC < 0.5 x 10^9/L) observed in chemotherapy cycle 1.

ELIGIBILITY:
Inclusion Criteria:

1. Show evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial.
2. Females ≥ 18 years of age and < 75 years of age.
3. Diagnosed with Stage II-IV breast cancer.
4. Subject is scheduled to undergo 4 cycles of TA chemotherapy (docetaxel, doxorubicin, 75, and 60 mg/m2, respectively).
5. ECOG Performance status of ≤ 2.
6. White Blood Cell count (WBC) ≥ 4.0 × 109/L, hemoglobin ≥ 11.5 g/dL and a platelet count ≥ 150 × 109/L.
7. Demonstrate adequate renal, hepatic function (Liver function tests (ALT, AST, alkaline phosphatase and total bilirubin)) should be less than 2.5x upper limits of normal (ULN). Serum creatinine should be less than 1.7x ULN.
8. All subjects must agree to use at least one of the following types of contraception: intrauterine device, implantable progesterone device, progesterone intramuscular injection, or oral contraceptive, which has been started at least one month prior to visit one and will continue for the duration of the trial. The contraceptive patch or condom use with spermicide is also acceptable forms of contraception as long as they will be used continually throughout the duration of the trial.

Exclusion Criteria:

1. Subject is <18 or ≥ 75 years of age.
2. Disease progression has occurred while receiving a taxane regimen.
3. Subject has undergone radiation therapy within 4 weeks of enrollment.
4. Subject has undergone bone marrow or stem-cell transplantation.
5. Subject has a history of prior malignancy other than breast cancer that is NOT in remission.
6. Subjects that have used G-CSF or any other drug that may potentiate the release of neutrophils (i.e. lithium) within 6 weeks of the screening period are excluded.
7. Subject has had chemotherapy within 365 days of screening.
8. Subject has documented congestive heart failure, cardiomyopathy or myocardial infarction by clinical diagnosis, ECG test, or any other relevant test.
9. History of alcohol or drug abuse that would interfere with the ability to be compliant with the study procedure.
10. Unwillingness to participate in the study.
11. Any underlying medical condition that, in the Investigator's opinion, would make the administration of study drug hazardous to the patient or that would obscure the interpretation of adverse events.
12. Receiving other investigational drugs or biologics within 1 month or five half lives of enrollment.
13. Any condition, which can cause splenomegaly.
14. Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease.
15. ALT, AST, alkaline phosphatase, total bilirubin ≥ 2.5 upper limit of normal.
16. Subject with active infection, or known to be infected with chronic active Hepatitis B within the last 1 year (unless shown at the time of study entry to be Hepatitis B antigen negative), or having any history of Hepatitis C.
17. Women who are pregnant or breast-feeding.
18. Subject known to be seropositive for HIV, or who have had an AIDS defining illness or a known immunodeficiency disorder.
19. Subject with a history of tuberculosis or exposure to tuberculosis. Patients that have received a prior chest X-ray for suspicion of tuberculosis are also excluded unless they have been confirmed to be PPD negative or they had latent tuberculosis that has been previously treated.
20. Subjects with Sickle Cell disease
21. Subjects with known hypersensitivity to E.coli derived proteins' pegfilgrastim' filgrastim, or any other component of the study drug.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin F Dreyer, Study Director — EVIVE Biotechnology
Locations (1):
- Covance, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glaspy J, Bondarenko I, Burdaeva O, Chen J, Rutty D, Li R, Wang S, Hou Q, Li S. Efbemalenograstim alfa, an Fc fusion protein, long-acting granulocyte-colony stimulating factor for reducing the risk of febrile neutropenia following chemotherapy: results of a phase III trial. Support Care Cancer. 2023 Dec 16;32(1):34. doi: 10.1007/s00520-023-08176-6. PMID 38103088

RESULTS

PARTICIPANT FLOW:
Period: Cycle 1
Arm/Group | F-627 | Placebo
Started | 83 | 39
Completed | 83 | 38
Not Completed | 0 | 1
Period: Cycle 2-4
Arm/Group | F-627 | Placebo
Started | 83 | 38 (1 subject withdrawn in Cycle 1)
Completed | 81 | 37
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | F-627 | Placebo | Total
Number analyzed (Participants) | 83 | 39 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (9.25) | 51.5 (9.00) | 51.0 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 39 | 122
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 82 | 38 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 82 | 39 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 0 | 1
  Ukraine | 46 | 22 | 68
  Russia | 32 | 16 | 48
  Hungary | 4 | 1 | 5
Reproductive Status [Count of Participants; unit: Participants]
  Childbearing potential | 37 | 15 | 52
  Non-childbearing potential - Post-menopausal | 42 | 23 | 65
  Non-childbearing potential - Surgically sterile | 4 | 1 | 5
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (5.36) | 27.4 (6.22) | 26.6 (5.65)
Baseline ECOG [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  Grade 0: fully active, able to carry on all pre-disease performance without restriction
  Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work
  Participants
    Grade 0 | 46 | 27 | 73
    Grade 1 | 37 | 12 | 49
Cancer Stage at Screening [Count of Participants; unit: Participants] — Doctors combine the tumor, node, metastasis results and other factors specific to cancer to determine the stage of cancer for each person. Most types of cancer have four stages: stages I to IV. Stage IV is considered a worse outcome than Stage I.
  Participants
    Stage II | 43 | 21 | 64
    Stage III | 22 | 12 | 34
    Stage IV | 18 | 6 | 24
Days from Diagnosis [Mean (Standard Deviation); unit: days] | 224.5 (572.21) | 445.9 (1337.99) | 294.6 (888.93)

OUTCOME MEASURES:

1. Primary Outcome: The Duration in Days of Grade 4 (Severe) Neutropenia Observed in Chemotherapy Cycle 1 in Comparison to Placebo
Description: Subjects will be randomized to F-627 or Placebo at 2:1 ratio. About 24 hours after chemotherapy, subjects will either receive 20mg fixed dose F-627 or Placebo. The subject's absolute neutrophil count (ANC) will be monitored each day post chemotherapy administration until the ANC level exceeds 2.0x10^9/L, then the value will be monitored every three days until the next chemotherapy cycle is entered. The duration of grade 4 neutropenia (ANC <0.5x10^9/L) in this cycle is the primary efficacy endpoint.
Time Frame: The first of 4, 21 Day Chemotherapy Cycles, an average of 3 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | Placebo
Number analyzed (Participants) | 83 | 39
days | 1.3 (1.17) | 3.9 (1.35)

2. Secondary Outcome: The Duration in Days of Grade 4 (Severe) Neutropenia (ANC < 0.5 × 10^9/L) for Chemotherapy Cycles 2, 3, and 4, and Over All Cycles.
Description: The duration of severe neutropenia will be measured for each patient during chemotherapy cycle 2-4 and over all cycles. Each chemotherapy is expected to last 21 days.
Time Frame: Over all 4 cycles, about 12 weeks
Population: Missing ANC data. No multiple imputation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | Placebo
Number analyzed (Participants) | 83 | 39
days
  Cycle 2: number analyzed (Participants) | 75 | 36
  Cycle 2 | 0.3 (0.76) | 0.8 (1.20)
  Cycle 3: number analyzed (Participants) | 72 | 32
  Cycle 3 | 0.3 (0.84) | 0.5 (1.19)
  Cycle 4: number analyzed (Participants) | 73 | 29
  Cycle 4 | 0.2 (0.62) | 0.7 (1.39)
  All cycles | 0.5 (0.62) | 1.4 (1.32)

3. Secondary Outcome: The Duration in Days of Grade 2 (Mild), Grade 3 (Moderate) and 4 (Severe) Neutropenia Over All Cycles.
Description: The duration in days of mild, moderate and severe neutropenia will be recorded for 4 chemotherapy cycles. Grade 2 neutropenia is when a patient's ANC<1.5x10^9/L, Grade 3 neutropenia is when a patient's ANC<1.0x10^9/L, and Grade 4 neutropenia is when a patient's ANC <0.5x10^9/L.
Time Frame: 4 chemotherapy cycles, about 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | Placebo
Number analyzed (Participants) | 83 | 39
days
  Grade 4 | 0.5 (0.62) | 1.4 (1.32)
  Grade 3 | 1.2 (1.08) | 1.9 (1.46)
  Grade 2 | 1.8 (1.24) | 2.7 (1.71)

4. Secondary Outcome: Number of Participants With Febrile Neutropenia (FN) for Each Chemotherapy Cycle and Over All Cycles
Description: Febrile neutropenia is defined as a single oral temperature of ≥38.3°C (101°F) or a temperature of >38.0°C (100.4°F) sustained for >1 hour and ANC < 0.5 x 10^9/L
Time Frame: 4 chemotherapy cycles, about 12 weeks
Population: 3 subjects terminated early.
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | Placebo
Number analyzed (Participants) | 83 | 39
Participants
  Cycle 1: Subjects with FN | 4 | 10
  Cycle 1: Subject without FN | 79 | 29
  Cycle 2: number analyzed (Participants) | 83 | 38
  Cycle 2: Subjects with FN | 0 | 1
  Cycle 2: Subject without FN | 83 | 37
  Cycle 3: number analyzed (Participants) | 82 | 37
  Cycle 3: Subjects with FN | 0 | 0
  Cycle 3: Subject without FN | 82 | 37
  Cycle 4: number analyzed (Participants) | 82 | 37
  Cycle 4: Subjects with FN | 0 | 0
  Cycle 4: Subject without FN | 82 | 37
  All cycles: Subjects with FN | 4 | 11
  All cycles: Subject without FN | 79 | 28

5. Secondary Outcome: Number of Participants With Grade 2, Grade 3, and Grade 4 Neutropenia for All Chemotherapy Cycles.
Description: The number of subjects with grade 2, 3 and 4 neutropenia will be recorded for all 4 chemotherapy cycles.
Time Frame: 4 chemotherapy cycles, about 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | Placebo
Number analyzed (Participants) | 83 | 39
Participants
  Grade 4 Neutropenia: yes | 58 | 37
  Grade 4 Neutropenia: no | 25 | 2
  Grade 3 Neutropenia: yes | 71 | 37
  Grade 3 Neutropenia: no | 12 | 2
  Grade 2 Neutropenia: yes | 77 | 37
  Grade 2 Neutropenia: no | 6 | 2

6. Secondary Outcome: The Time in Days to ANC Recovery Post Nadir for Each Chemotherapy Cycle and Over All Cycles; Recovery Defined as an ANC ≥ 2.0 × 10^9/L After the Expected ANC Nadir.
Description: The time to ANC recovery post nadir for each patient, for each of their chemotherapy cycles will be recorded. Recovery for this protocol is defined as achieving an ANC ≥ 2.0 × 10^9/L after the expected ANC nadir (expected nadir is typically 4-6 days post chemotherapy administration).
Time Frame: 4 chemotherapy cycles, about 12 weeks
Population: 3 Subjects terminated early (1 in F-627 arm, 2 in the placebo arm). In addition, 1 subject in placebo arm reached her Nadir(1.81) at Day 7 but the rest of ANC values are missing. Because the recovery information is not available, this subject was removed from the Time to ANC recovery analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | Placebo
Number analyzed (Participants) | 83 | 39
days
  Cycle 1: number analyzed (Participants) | 83 | 38
  Cycle 1 | 2.1 (1.08) | 4.0 (2.07)
  Cycle 2: number analyzed (Participants) | 83 | 38
  Cycle 2 | 1.6 (1.35) | 2.0 (1.37)
  Cycle 3: number analyzed (Participants) | 82 | 37
  Cycle 3 | 1.6 (1.34) | 1.7 (1.79)
  Cycle 4: number analyzed (Participants) | 82 | 36
  Cycle 4 | 1.9 (1.39) | 1.5 (1.73)
  All cycles | 1.8 (0.94) | 2.4 (1.20)

7. Secondary Outcome: The Depth of the ANC Nadir for Each Chemotherapy Cycle and Over All Cycles.
Description: The depth of ANC nadir for each cycle is the minimal ANC value (× 10^9/L ) for a patient in each chemotherapy cycle
Time Frame: 4 chemotherapy cycles, about 12 weeks
Population: 3 subjects terminated early.
Measure: Mean (Standard Deviation); unit: cells/10^9/L
Arm/Group | F-627 | Placebo
Number analyzed (Participants) | 83 | 39
cells/10^9/L
  Cycle 1 | 0.7 (1.16) | 0.2 (0.57)
  Cycle 2: number analyzed (Participants) | 83 | 38
  Cycle 2 | 2.0 (1.71) | 1.6 (1.71)
  Cycle 3: number analyzed (Participants) | 82 | 37
  Cycle 3 | 1.7 (1.58) | 1.8 (1.63)
  Cycle 4: number analyzed (Participants) | 82 | 37
  Cycle 4 | 1.7 (1.45) | 2.3 (2.01)
  All cycles | 1.5 (1.20) | 1.4 (1.23)

8. Secondary Outcome: Number of Participants With Infections for Each Chemotherapy Cycle and Over All Cycles.
Description: The number of subjects with infections for each arm of the study will be recorded for each and all 4 chemotherapy cycles.
Time Frame: 4 chemotherapy cycles, about 12 weeks
Population: Some subjects terminated earlier
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | Placebo
Number analyzed (Participants) | 83 | 39
Participants
  Cycle 1: Subjects with infection | 2 | 3
  Cycle 1: Subjects without infection | 81 | 36
  Cycle 2: number analyzed (Participants) | 83 | 38
  Cycle 2: Subjects with infection | 1 | 2
  Cycle 2: Subjects without infection | 82 | 36
  Cycle 3: number analyzed (Participants) | 82 | 37
  Cycle 3: Subjects with infection | 5 | 3
  Cycle 3: Subjects without infection | 77 | 34
  Cycle 4: number analyzed (Participants) | 82 | 37
  Cycle 4: Subjects with infection | 1 | 0
  Cycle 4: Subjects without infection | 81 | 37
  All cycles: Subjects with infection | 9 | 8
  All cycles: Subjects without infection | 74 | 31

9. Secondary Outcome: Number of Participants With Use of Antibiotics and Pain Medications
Description: Antibiotics and pain medications use will be recorded for each chemotherapy cycle and overall cycles
Time Frame: 4 chemotherapy cycles, about 12 weeks
Population: 3 subjects terminated early
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | Placebo
Number analyzed (Participants) | 83 | 39
Participants
  Cycle 1: antibiotic and pain medications use | 9 | 13
  Cycle 1: no antibiotic and pain medications use | 74 | 26
  Cycle 2: number analyzed (Participants) | 83 | 38
  Cycle 2: antibiotic and pain medications use | 3 | 2
  Cycle 2: no antibiotic and pain medications use | 80 | 36
  Cycle 3: number analyzed (Participants) | 82 | 37
  Cycle 3: antibiotic and pain medications use | 2 | 1
  Cycle 3: no antibiotic and pain medications use | 80 | 36
  Cycle 4: number analyzed (Participants) | 82 | 37
  Cycle 4: antibiotic and pain medications use | 1 | 0
  Cycle 4: no antibiotic and pain medications use | 81 | 37
  All cycles: antibiotic and pain medications use | 13 | 15
  All cycles: no antibiotic and pain medications use | 70 | 24

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the time of randomization until 28 days after completion of the trial (a total of 16 weeks) or 28 days after premature withdrawal of a subject from the trial.
Groups:
- Cycle 1 F-627; All 4 Cycles F-627: F-627, 20 mg fixed dose pre-filled syringe, dosed Day 2 of each of 4 chemotherapy cycles.
- Cycle 1 Placebo: Placebo, pre-filled syringe administered Day 2 of the first chemotherapy cycle 1
- Cycle 1 Placebo and Cycle 2-4 F-627: Placebo, pre-filled syringe administered Day 2 of the first chemotherapy cycle; and F-627, 20 mg fixed dose pre-filled syringe administered Day 2 of each of the following 3 chemotherapy cycles.
Arm/Group | Cycle 1 F-627 | Cycle 1 Placebo | All 4 Cycles F-627 | Cycle 1 Placebo and Cycle 2-4 F-627
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/39 | 0/83 | 0/39
Serious Adverse Events (participants affected / at risk) | 4/83 | 10/39 | 4/83 | 11/39
Other Adverse Events (participants affected / at risk) | 17/83 | 5/39 | 26/83 | 9/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 1 F-627 (N=83) | Cycle 1 Placebo (N=39) | All 4 Cycles F-627 (N=83) | Cycle 1 Placebo and Cycle 2-4 F-627 (N=39)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 10 | 3 | 11
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 1 F-627 (N=83) | Cycle 1 Placebo (N=39) | All 4 Cycles F-627 (N=83) | Cycle 1 Placebo and Cycle 2-4 F-627 (N=39)
Nausea (Gastrointestinal disorders) | 6 | 1 | 8 | 3
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 5 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 2 | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 5 | 1
Fatigue (General disorders) | 3 | 2 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT02872103/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT02872103/SAP_002.pdf